CLINICAL TRIAL: NCT03893422
Title: An Placebo-Controlled Clinical Nutrition Study to Evaluate the Metabolic Effects of Two Medical Food Products in Subjects With Type 2 Diabetes Treated With Diet and Exercise Alone or in Combination With Metformin ± Sulfonylurea
Brief Title: Placebo-Controlled Clinical Nutrition Study of the Safety and Metabolic Effects of Two Medical Foods in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pendulum Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: WB201-202
Record Dates: First submitted 2019-03-13; First posted 2019-03-28 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: glucose control; inflammation; safety; microbiome
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Inflammation

STUDY DESIGN:
Intervention Model Description: Balanced randomization across 3 arms: formulation WB-010, formulation WB-011 and placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study product was provided for each arm in identical capsules
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- WB-010 (Experimental): 3 capsules administered twice daily with morning and evening meal for 12 weeks
  Interventions: Other: WB-010
- WB-011 (Experimental): 3 capsules administered twice daily with morning and evening meal for 12 weeks
  Interventions: Other: WB-011
- Placebo (Placebo Comparator): 3 capsules administered twice daily with morning and evening meal for 12 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Other: WB-010 — Medical food formulation
  Arms: WB-010
Other: WB-011 — WB-011 medical food product
  Arms: WB-011
Other: Placebo — Placebo Capsules identical to those containing WB-010 and WB-011.
  Arms: Placebo

SUMMARY:
This 16 week placebo-controlled study evaluates the safety and impact of two medical food study products, WBF10 and WBF11, consisting of commensal microbes. The primary endpoints were safety, glucose AUC during meal tolerance test and C reactive protein (CRP)..

DETAILED DESCRIPTION:
Targeting the microbiome for treating metabolic syndrome has been gaining traction with multiple population studies demonstrating a difference between healthy individuals and patients with metabolic syndrome. Whole Biome has identified and created two medical food formulations (MFFs) aimed at improving metabolic syndrome via two mechanisms of action targeting the microbiome: (1) increasing butyrate production and (2) increasing mucin regulation.

This randomized, parallel-group, placebo-controlled, double-blinded study assesses the safety and metabolic effects of 2 MFFs on glucose control and the generalized inflammatory state associated with Type 2 Diabetes. The microbes have been fully characterized, certified as Generally Recognized As Safe (GRAS) and manufactured to Good Manufacturing Practice (GMP) standards. The target population was patients with Type 2 Diabetes who either had not been treated with antidiabetic agents or treated with metformin +/- a sulfonylurea. Subjects were randomized in a balanced manner to receive capsules containing placebo, WBF10 or WBF11.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes treated with diet and exercise alone or in combination with metformin and/or sulfonylurea
* If treated with metformin and/or sulfonylurea, must have been on a stable dose of the drug(s) for a minimum of 3 months with a stable A1c value
* If treated with diet and exercise alone, must have one of the following:

  * Documented fasting plasma glucose >126 mg/dL
  * A1c value ≥6.8%
* If treated with diet and exercise + metformin and/or sulfonylurea, must have a stable A1c between 6.8% and 11.0% for 3 months prior study entry
* BMI >25 but <45 and weight stable within +/- 5% over past 3 months
* If female, must meet all the following criteria:

  * Not pregnant or breastfeeding
  * If of childbearing potential (including peri-menopausal women with menstruation during past year) must practice and be willing to continue appropriate birth control during the entire duration of the study
* Have a home freezer available for immediate freezing of stool samples
* Able to read, understand, and sign the informed consent form (ICF) and HIPAA authorization when applicable,
* Able to communicate with the investigator, and understand and comply with protocol requirements

Exclusion Criteria:

* Use of antibiotic, antifungal, antiparasitic, or antiviral therapy within 30 days prior to study entry
* Planned use or antibiotic, antifungal, antiparasitic, or antiviral treatment during the study period
* Subjects using a proton pump inhibitor must be on a stable dose that will be maintained throughout the study period
* Present use of probiotics/nutritional supplements. (Note: Use of replacement doses of Vitamin D, calcium supplements, and a single daily multi-vitamin tablet allowed)
* Participation in a structured weight-loss program within the past 2 months
* Change in body weight ≥5% within the past month
* Excess alcohol consumption; with an alcoholic drink defined as 12 fluid ounces of beer (5% alcohol), 5 fluid ounces of wine (12% alcohol) or 1.5 fluid ounces of 80 proof distilled spirits

  * Women: More than 2 alcoholic drinks/day or more than 7 drinks/week
  * Men: More than 3 alcoholic drinks/day or more than 10 drinks/week
* Travel outside United States within 30 days of study entry
* Planned travel outside United States during study period
* Use of an experimental drug within 30 days prior to study entry
* Known milk, peanut, tree nut, wheat, soy or shellfish allergy
* Diagnosis of a sexually transmitted disease including, but not limited to, HIV, syphilis, herpes, gonorrhea, hepatitis A, hepatitis B, and hepatitis C
* Hospitalization during last 3 months (Same day surgery center procedures allowed)
* Active GI disease
* Gastrointestinal tract surgery (appendectomy and cholecystectomy allowed)
* Cystic fibrosis
* Any condition deemed by the investigator to disqualify subject

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2017-10-22 (Actual); Primary Completion 2018-08-16 (Actual); Study Completion 2018-09-14 (Actual)

PRIMARY OUTCOMES:
3-hour plasma glucose AUC | From Baseline to Week 12
  Change in area under plasma glucose concentration versus time curve (AUC) during standardized 3-hour Meal Tolerance Test
CRP | From Baseline to Week 12
  Change in c-reactive protein concentration

SECONDARY OUTCOMES:
Incremental glucose AUC | From Baseline to Week 12
  Change in area under plasma glucose concentration versus time curve (AUC) above the fasting plasma glucose level during standardized 3-hour Meal Tolerance Test
Hemoglobin A1c | From Baseline to Week 4 and Week 12
  Change in A1c
Fasting plasma glucose concentration | From Baseline to Weeks 4, 8 and 12
  Change in fasting plasma glucose concentration
Fasting plasma insulin concentration | Baseline to Weeks 4, 8 and 12
  Change in fasting plasma insulin concentration
Plasma insulin AUC | From Baseline to Week 12
  Change in area under plasma insulin concentration versus time curve (AUC) during standardized 3-hour Meal Tolerance Test
Homeostatic Model Assessment (HOMA) of Insulin Resistance (IR) | From Baseline to Week 12
  Change in HOMA-IR
Matsuda index | From Baseline to Week 12
  Change in Matsuda index
Fasting Lipid Panel | From Baseline to Week 12
  Change in fasting serum concentrations of total cholesterol, LDL cholesterol, HDL cholesterol and triglycerides
Inflammatory markers | From Baseline to Week 12
  Change in concentrations of interleukin-6, interleukin-10, tumor growth factor-α and T-cell growth factor-beta
Body weight in kilograms | From Baseline to Weeks 2, 4, 8 and 12
  Change in body weight in kilograms
Body Mass Index (BMI) | At Baseline
  BMI = weight in kg/m2
Waist Circumference | From Baseline to Weeks 2, 4, 8 and 12
  Change in Waist Circumference
Fecal Microbiome Profile | From Baseline to Week 12
  Change in Fecal Microbiome Profile assessed by DNA sequencing
Adverse Events | From Baseline to Week 12
  Number of participants with adverse events related to therapy
Laboratory (Chemistry panel + CBC) Values | From Baseline to Week 12
  Number of Participants With Abnormal Laboratory Values Related to Therapy
Hospital Anxiety and Depression Scale | From Baseline to Week 12
  Subjects respond to 14 questions; 7 anxiety focused and 7 depression focused. Responses of "not at all", "not much", "sometimes" and "definitely" are translated to a numerical score of 0 to 4 respectively. For 2 of the depression related questions, the scoring scale is reversed. The individual numerical scores are added to provide an overall score which is interpreted as follows: 0 to 7 graded a non-case, 8 to 10 graded a borderline case and 11+ graded a case. An increase in the overall numerical score from baseline to Week 12 represents worsening and a decrease in the numerical score from baseline to Week 12 represents improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Orville G Kolterman, MD, Principal Investigator — Pendulum Therapeutics
Locations (5):
- United States (5):
  - Science 37, Torrance, California
  - Orange County Research Center, Tustin, California
  - Northside Medical Center, Youngstown, Ohio
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Juno Research, LLC, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Perraudeau F, McMurdie P, Bullard J, Cheng A, Cutcliffe C, Deo A, Eid J, Gines J, Iyer M, Justice N, Loo WT, Nemchek M, Schicklberger M, Souza M, Stoneburner B, Tyagi S, Kolterman O. Improvements to postprandial glucose control in subjects with type 2 diabetes: a multicenter, double blind, randomized placebo-controlled trial of a novel probiotic formulation. BMJ Open Diabetes Res Care. 2020 Jul;8(1):e001319. doi: 10.1136/bmjdrc-2020-001319. PMID 32675291